CLINICAL TRIAL: NCT03550690
Title: The Quality of Life of Patients Who Have Rocket Indwelling Pleural Catheter Drainage or Repeated Large Volume Paracentesis - Observational Feasibility Study
Brief Title: Quality of Life of Patients Who Have Rocket Indwelling Pleural Catheter Drainage or Repeated Large Volume Paracentesis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gloucestershire Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Paul Perkins, Consultant in Palliative Medicine, Gloucestershire Hospitals NHS Foundation Trust
Other Study IDs: Rocket Project 1; 242415 (Other: IRAS)
Record Dates: First submitted 2018-05-26; First posted 2018-06-08 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Ascites, Malignant
MeSH Terms: conditions — Ascites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Large Volume Paracentesis: Patient has repeated large volume paracentesis for recurrent ascites secondary to cancer
  Interventions: Device: Large Volume Paracentesis
- Semi-permanent drain: Patient has a semi-permanent drain (Rocket Indwelling Pleural Catheter) placed for recurrent ascites secondary to cancer
  Interventions: Device: Rocket Indwelling Pleural Catheter

INTERVENTIONS:
Device: Large Volume Paracentesis — Insertion of a plastic tube into the abdomen and draining off ascitic fluid under local anaesthetic, removing the drain afterwards
  Groups: Large Volume Paracentesis
Device: Rocket Indwelling Pleural Catheter — A small plastic tube under the skin which is left in place so that the fluid can be drained if it builds up again
  Groups: Semi-permanent drain

SUMMARY:
Ascites (accumulation of fluid in the abdominal cavity) is a common problem which can lead to distressing symptoms. When caused by cancer, management options are chemotherapy, diuretics and ascitic drainage. Ascitic drainage is performed by inserting a plastic tube into the abdomen and draining off the fluid under local anaesthetic, removing the drain afterwards. For some, the fluid will return and the procedure needs repeating. A relatively new treatment involves inserting a semi-permanent drain - a small plastic tube under the skin which is left in place so that the fluid can be drained if it builds up again. The potential benefit to patients is that afterwards they can have fluid removed at home. This might reduce the number of hospital admissions, outpatient visits and the number of procedures they need to have in the last few months of life. In Gloucestershire, the Rocket Indwelling Pleural Catheter (IPC) is the semi-permanent drain of choice.

Our research group has a particular interest in the management of ascites and we recently completed the first qualitative interview study with patients with this condition - patients with ascites secondary to cancer. Patients were pleased to have semi-permanent drains in place as it meant that repeated admissions to hospital were avoided. They did not have to wait for a build-up of fluid before more could be drained off; and symptoms never had to build up as badly as when they were having repeated ascitic drainage.

We plan a feasibility study to ascertain whether a definitive non-randomised study to detect differences in quality of life between Rocket IPC and repeat ascitic drainage is possible and how many patients would be needed for such a study.

DETAILED DESCRIPTION:
Study Objective This feasibility study aims to establish how best to conduct a definitive prospective non-randomised QOL study for patients with malignant ascites who either have placement of a Rocket IPC or repeated LVP

Study Design This is an open label, non-randomised observational study. Each patient will receive verbal and written information followed by signing of an Informed Consent Form prior to participation. They will be asked to capture data about their QOL by completing paper diaries.

If the patient has a relative / next of kin we will ask permission from the patient to approach them to see if they would be happy to consent to helping with data collection for the study.

Study Procedures

When patients are booked for ascitic drainage in hospitals or hospice a member of the patient's clinical team will discuss the study with the patient (either in person or via telephone). If in agreement, the doctor / nurse will pass on their contact details to a member of the research team who will then telephone the patient and:

* Ask the patient if they would be happy to receive a patient information leaflet by post or email
* Ask the patient if they would be happy for their relative / next of kin to be contacted about this study. The relative / next of kin will then be contacted and, if they are happy to receive it, a participant information leaflet will be posted or emailed to them.

[If the patient is having an IPC fitted the relative may fit the inclusion criteria for the related study, Rocket Project 2, so that this study may be discussed at this point and a participant information leaflet provided too.]

At the time of admission for the procedure informed consent will be obtained from the patient and the following information will be obtained and recorded on a case report form:

* Patient's age, gender, diagnosis
* Performance status
* How many LVPs the patient has had up until the current procedure
* Patient's understanding of treatment options for ascites management, in particular whether Rocket IPC has been mentioned
* Why was this option chosen?
* Opinion about participation in a randomised trial if one was being conducted The research nurse will ensure that baseline blood tests to include renal function and albumin have been performed prior to the procedure.

Rarely, a patient could be referred for the procedure and have it performed later that day. In that scenario we would like to have permission for a cooling off period to be waived by the participants - we would argue that this is not a particularly burdensome study.

Informed consent will also be sought from the relative / next of kin. It will usually be possible to do obtain this when the patient attends for the procedure but a separate appointment to obtain informed consent may be needed at the relative / next of kin's home or care setting.

A patient can be recruited to the study if their relative / next of kin does not consent OR they have no relative / next of kin.

A four week diary will be given to the patient to capture the following information:

1. Number of LVPs / Rocket IPC drainage episodes performed*
2. Volumes of fluid removed at LVPs OR number of Rocket IPC bottles used at Rocket IPC drainage*
3. Any complications - catheter blockage, infections, hospital admissions*
4. The Edmonton Symptom Assessment System:Ascites Modification (ESAS:AM) DAILY
5. The EuroQol questionnaire (EQ-5D) as a generic QOL measure DAILY
6. The European Organization for the Research and Treatment of Cancer (EORTC) Core QOL Questionnaire (QLQ-C30) WEEKLY
7. Anti-cancer treatment received by the patient*
8. Diuretics received by the patient*

If a relative / next of kin has consented they can help the patient to complete their diary. They will not be able to give a proxy measure for any of the quality of life scores but will be able to assist the patient with completion of these and also with objective measures (e.g. those marked * above) The research nurse will contact the patient frequently by phone, to provide support with data collection, if required.

When the patient is close to completing 4 weeks in the study they will be offered the opportunity to complete another 4 week diary. It will be explained to them that this is not essential but will provide useful information.

When close to completing the 2nd 4 week diary (i.e. after 8 weeks) they will, once again, be offered a further diary. Patients will complete a maximum of three diaries.

Patients will not be expected to complete questionnaires if they do not feel well enough or lose capacity. Patients' clinical course can fluctuate and there may be a time when they feel well enough to complete questionnaires again. Data about fluid volumes removed may still be collected after a patient loses capacity by healthcare staff, as is routine practice, or consenting relatives / next of kin.

Only patients with capacity will be approached for participation in the study.

Blood Tests Renal function and albumin will be measured at baseline, 6 weeks and 12 weeks (the latter 2 time points only if the patient remains in the study after 4 weeks and 8 weeks) - if necessary performed by the research nurse at patient's home.

Blood tests will not be performed on patients who have lost capacity for the purposes of this study. If patients without capacity have blood tests taken for other reasons the results will be used as part of data analysis.

Only a very small percentage of people living in Gloucestershire are not English speaking. It has been decided that it is not cost effective to fund translation for this feasibility study. The information on the numbers of patients / carers who may have been excluded and the languages that might have been needed will be collected and this will be taken into account when planning a larger study.

Outcome measures

There have been recommendations about suitable QOL measures for use with patients with ascites. We discussed these with service users and carers and have agreed on using for this study:

1. The Edmonton Symptom Assessment System:Ascites Modification (ESAS:AM)
2. The EuroQol questionnaire (EQ-5D) as a generic QOL measure
3. The European Organization for the Research and Treatment of Cancer (EORTC) Core QOL Questionnaire (QLQ-C30)

In addition we will ask healthcare professionals, patients or consenting carers (depending on who manages the drain) to record volumes of fluid removed at each paracentesis and episode of semi-permanent drainage.

We will ask patients and carers about:

Drainage complications and hospital admissions. Chemotherapy use Diuretic use

Withdrawal of subjects from the study

Patients will cease participation in the study when one of the following criteria is met:

They choose to withdraw They choose not to complete a further QOL diary They complete their third monthly QOL diary They lose capacity and it is thought that this will be permanent

Carers will cease participation in the study when one of the following criteria is met:

They choose to withdraw The patient dies

A patient may remain in the study although a carer / next of kin has withdrawn and vice versa.

Statistical Analysis Percentage presence and percentage completeness of the three QOL measures will be evaluated. These results will allow an estimation of the number of patients, resources and time needed to perform a definitive prospective non-randomised QOL study for patients with malignant ascites who either have placement of a Rocket IPC or repeated LVP.

The following analysis will also be conducted:

* QLQ-C30 and EQ-5D averaged for each participant for the duration of their participation, using the area under the curve method.
* ESAS:AM analysed by estimating the prevalence of individual symptoms at each time point, as well as the time-weighted average burden of symptoms for each participant.

It is hoped that data from the feasibility study can be used in the definitive study if the methodology of the two studies remains the same.

We estimate over a 6-month period approximately 60 patients with ascites secondary to cancer will have a paracentesis. We plan to recruit 20 patients having a drainage procedure (LVP or Rocket IPC) within 6 months.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Male or female adult patients
2. Have ascites due to cancer undergoing treatment at Gloucestershire Hospitals NHS Foundation Trust
3. Planned to have an ascitic tap within a week
4. Thought to have an estimated prognosis of 12 weeks or more
5. Willing and able to provide signed written informed consent

Patient Exclusion Criteria

1. Patients who, in the opinion of the clinical team, would be too distressed by the idea of participation.
2. Patients who might not adequately understand verbal explanations or written information given in English.

Relative Inclusion Criteria:

1. Adult supporting patient participant in Rocket Project 1
2. Happy to support patient with completion of patient diaries

Relative Exclusion Criteria

1. Relatives who, in the opinion of the clinical team, would be too distressed by the idea of participation.
2. Relatives who might not adequately understand verbal explanations or written information given in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See above
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Percentage presence and percentage completeness of the three QOL measures | 3 months

SECONDARY OUTCOMES:
Number of LVPs / Rocket IPC drainage episodes performed | 3 months
Volumes of fluid removed at LVPs OR number of Rocket IPC bottles used at Rocket IPC drainage | 3 months
Complications | 3 months
  Catheter blockage, infections, hospital admissions
The Edmonton Symptom Assessment System:Ascites Modification (ESAS:AM) DAILY | 3 months
The EuroQol questionnaire (EQ-5D) as a generic QOL measure DAILY | 3 months
The European Organization for the Research and Treatment of Cancer (EORTC) Core QOL Questionnaire (QLQ-C30) WEEKLY | 3 months
Anti-cancer treatment received by the patient | 3 months
Diuretics received by the patient | 3 months

IPD SHARING:
Plan to Share IPD: No
Available on request

REFERENCES:
- [Background] Day R, Mitchell T, Keen A, Perkins P. The experiences of patients with ascites secondary to cancer: a qualitative study. Palliat Med. 2013 Sep;27(8):739-46. doi: 10.1177/0269216313480400. Epub 2013 Apr 4. PMID 23558342
- [Background] Easson AM, Bezjak A, Ross S, Wright JG. The ability of existing questionnaires to measure symptom change after paracentesis for symptomatic ascites. Ann Surg Oncol. 2007 Aug;14(8):2348-57. doi: 10.1245/s10434-007-9370-3. Epub 2007 May 16. PMID 17505860